CLINICAL TRIAL: NCT02260765
Title: Post Marketing Study to Evaluate the Resource Utilization of Patients Suffering From Resistant Depression Treated With Deep TMS in Comparison to Treatment as Usual
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was never funded therefore no patients were enrolled.
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HCP-Post Marketing-Brainsway
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Depression
Keywords: Treatment as Usual = TAU
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCP dTMS (Active Comparator): this arm will receive dTMS treatment
  Interventions: Device: dTMS
- HCP TAU (No Intervention): this arm will continue with the same drugs that they are using usually, which mean treatment as usual

INTERVENTIONS:
Device: dTMS — The Brainsway H-Coil TMS device is intended for the treatment of depressive episodes in patients suffering from Major Depressive Disorder (MDD). The device technology is based on the application of deep TMS by means of repetitive pulse trains at a determined frequency
  Arms: HCP dTMS

SUMMARY:
The aim of the study is to evaluate the efficacy of the Deep TMS compare to TAU and the different in resource utilization of treating depression with Deep TMS compare to the TAU.

The current study is a prospective semi-naturalistic, randomized study in which depressed patient who failed to respond to at least one medication or could not tolerate at least two antidepressants and are seeking for alternative treatment will be offered to join an open label study. The study designed as double arm study of which patient will have 50% chance to be randomized to one of the study groups.

The study includes two arms. The dTMS study group will be treated according to the cleared FDA treatment protocol of 4 weeks of daily treatment following by additional 12 weeks of biweekly treatment and overall of 44 treatments. The Treatment As Usual arm will be treated by their primary care physician / psychiatrist according to the usual treatment recommend to the patient clinical status

DETAILED DESCRIPTION:
many patients do not respond to antidepressant or could not tolerate the adverse events. Hence, many patients are looking for medical alternatives. Those alternatives include psychotherapy, ECT, and TMS. The direct cost of those treatments is relatively high compare to antidepressants. However, the indirect costs including hospitalizations, physician visit, ER visits, pharmacy claims, labs and adverse events management may increase the overall costs and burden of illness for the health system. This study aims to evaluate the efficacy of the Deep TMS compare to TAU and the different in indirect costs of treating depression with Deep TMS compare to the TAU.

The current study is a prospective semi-naturalistic, randomized study in which depressed patient who failed to respond to at least one medication or couldn't tolerate at least two antidepressants and are seeking for alternative treatment will be offered to join an open label study. Patients eligible for the study will be asked to sign the informed consent. Than patients will be randomized to either Deep TMS treatment or TAU. The Deep TMS study group will receive the TMS treatment protocol as was cleared by the FDA. The TAU study group will be treated by their primary care physician / psychiatrist according to the usual treatment recommend to the patient's clinical status. Patient may continue its current treatment (with / without medications) or switch to a new treatment. However, treatment should be stable for at least 30 days prior to baseline visit except of Fluoxetine in which 45 days are required. Patients will be followed at 4 weeks and 6 month following baseline visit. The deep TMS treatment includes 4 weeks of acute daily treatment (20 treatments) following by 12 weeks of biweekly maintenance treatment. The purpose of the study is to explore the efficacy of the Deep TMS treatment compare to TAU and to investigate the differences in resource utilization between the study groups. The study population will be based on the FDA cleared patient population for the Deep TMS treatment. Safety will be assessed by monitoring of adverse events Other assessment scales will be used during the course of the study. Efficacy will be assessed using the Hamilton Depression Rating Score (HDRS), the self-reported questionnaires the QIDS-SR and the PHQ-9. Quality of life will be assessed by the Q-Les-Q questionnaire. Disability will be assessed by the Sheehan Disability Scale.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Patients at Healthcare Partners for at least one year
* Men and women 22-68 years of age
* Primary DSM-IV diagnosis of Major Depression, single or recurrent episode confirmed in Health Care Partners (HCP) database by ICD-9 diagnosis code
* Subject with QIDS score > 14 Subject with an HDRS-21 score > 22
* If treating with antidepressants patient should be stable on treatment for at least 30 days prior to baseline visit or 45 days in case of Fluoxetine
* Capable and willing to provide informed consent
* Able to adhere to the treatment schedule

Exclusion Criteria:

* QIDS-SR item 12 " Thoughts of Death or Suicide " score ≥3 or HDRS- 21 item 3 "Suicidal Ideation" score ≥3
* Depression secondary to a general medical condition, or substance- induced;
* History of substance abuse or dependence within the past 6 month (except nicotine and caffeine)
* Schizophrenic disorder
* Schizoaffective disorder
* Bipolar disorder, except when mania/hypomania was related to administration of antidepressant medications
* Major depression with psychotic features in the current episode
* Delusional disorder (current or within the past year)
* Eating disorders (current or within the past year)
* Obsessive compulsive disorder (current or within the past year)
* Post-traumatic stress disorder (current or within the past year)
* Current (or within 12 months of baseline) generalized anxiety disorder, panic disorder or social anxiety disorder as assessed by the investigator to be primary, causing a higher degree of distress or impairment than MDD.
* Current (or within 12 months of baseline) personality disorder (such as antisocial, schizotypal, histrionic, borderline, narcissistic) as assessed by the investigator to be primary, causing a higher degree of distress or impairment than MDD.
* Patients who have conductive, ferromagnetic or other magnetic- sensitive metals implanted in their head or within 30 cm of the treatment coil. Examples include cochlear implants, implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewelry and hair barrettes
* Patients who have active or inactive implants (including device leads), including cardiac pacemakers, implanted defibrillators, deep brain stimulators, cochlear implants, and vagus nerve stimulators
* Known or suspected pregnancy
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse
* Minimal MT found for both hands is higher than 70% of stimulator power output

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
HDRS-21 | Baseline and after 4 week from the baseline
  The primary efficacy endpoint is the change from baseline to 4 weeks visit in HDRS-21 score The change in HDRS-21 from baseline to 4 weeks visit will be compared between the treatment groups using a repeated measures analysis of covariance (ANCOVA, SAS® MIXED procedure). Baseline HDRS-21, antidepressant treatment at baseline, will be used as covariates. Baseline HDRS-21 scores and antidepressant treatment at baseline will be entered as continuous variables so that the potential for co-linearity problems will be minimized. Remission is defined as HDRS-21 score < 10. The remission rates at week 4 in the two groups will be compared using the Chi-square test or Fisher's exact test, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Alexander Bystritsky, MD, PhD, Principal Investigator — Healthcare Partners
Locations (1):
- Healthcare Partners, Los Angeles, California, United States